CLINICAL TRIAL: NCT07067983
Title: Clinical Evaluation of GRAPE Model for Gastric Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Professor, Zhejiang Cancer Hospital
Other Study IDs: IIT-2025-160
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Results following systematic screening — The GRAPE model's output (positive or negative) determines whether patients require follow-up gastroscopy

SUMMARY:
A Prospective Study Evaluating the Performance of the GRAPE Model in Gastric Cancer Screening and Its Detection Rates Across Different Disease Stages

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* Individuals undergoing thoracoabdominal CT examination
* Voluntarily participated in the study and provided written informed consent

Exclusion Criteria:

* Patients with confirmed diagnosis of gastric cancer
* Individuals with severe intellectual disabilities or communication disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing thoracoabdominal CT examination
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
GRAPE systematic screening results | first visited at baseline
  Screen-positive individuals after GRAPE systematic screening

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No